CLINICAL TRIAL: NCT04669834
Title: Effect of Core Stability Exercise on Temporal Activation of Core Muscles and Vasti in Isolated Patellofemoral Osteoarthritis.
Brief Title: Effect of Core Stability Exercise on Isolated Patellofemoral Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jilan Adel yousef, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: (P.T.Rec/012/002987)
Record Dates: First submitted 2020-12-02; First posted 2020-12-17 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Chondromalacia Patellae
MeSH Terms: conditions — Chondromalacia Patellae

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into two groups, group A and group B . Patients in both groups will receive a traditional physical therapy treatment, but group (B) will receive additional core stability exercise.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Other): Patients in this group will receive a traditional therapeutic knee rehabilitation program based on a recent systematic review in the form of mini-squatting exercise (up to 45 degree knee flexion measured by a universal goniometer) , strengthening of hip abductors and external rotators using clamshell exercise . No emphasis will be placed on stabilizing the core musculature before initiating any of those exercises.
  Interventions: Other: a traditional therapeutic knee rehabilitation program
- group B (Experimental): Patients in this group will receive the same program as group (A) plus core stability exercise , but the principles of core stability will be explained to patients before initiation of treatment and patients will be asked to comply with these principles during exercise. These principles include learning how to activate transversus abdominus by abdominal bracing without allowing pelvis tilting and ensure neutral spine and diaphragmatic breathing during exercise.
  Interventions: Other: a traditional therapeutic knee rehabilitation program; Other: core stability exercise

INTERVENTIONS:
Other: a traditional therapeutic knee rehabilitation program — mini-squatting exercise and clamshell exercise
Other: core stability exercise — the principles of core stability will be explained to patients before initiation of treatment and patients will be asked to comply with these principles during exercise. These principles include learning how to activate transversus abdominus by abdominal bracing without allowing pelvis tilting and ensure neutral spine and diaphragmatic breathing during exercise.
  Arms: group B

SUMMARY:
Purpose: to investigate the effect of core stability on PF OA. Methods: Thirty-one females with PF OA will be recruited. Patients will be randomly assigned into two groups, group A and group B . Patients in both groups will receive a traditional physical therapy treatment, but group (B) will receive additional core stability exercise. All patients will be evaluated for pain, functional performance, and muscular recruitment strategies (onset and duration) of multifidus, transversus abdominus (TrA), gluteus medius (GM), and vasti measured by quantitative Electromyography during stair ascent. pre and post-treatment.

DETAILED DESCRIPTION:
A) Procedures for evaluation:

The practical section of the studywill be undertaken in 6 weeks (2 sessions a week). Measurement will be taken before the start of treatment program then after the end of 6 weeks treatment program f in the following manner:

1. Patients will be asked to respond to the questions of the Kujala scale.
2. The eleven-point numerical rating scale will be used to measure pain severity
3. Investigators will collect the EMG activity of VMO, VL, GM, multifidus, and TrA using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels highresolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).

   Electromyographic data will be sampled at 1000 Hz and bandpass filtered at 50-200 Hz. For each muscle, three electrodes will be used; two electrodes will be placed ~ 30 mm apart in the direction of the muscle fibers and a ground electrode will be placed over the closest bony prominence. Before placement of the electrodes, the subject's skin will be cleaned with alcohol to reduce impedance and excess hair will be removed to eliminate shifting of the electrodes if needed. The stair-stepping task will consist of ascending 2 steps (each step will be 40 cm in width, 20 cm in height, without handrails. The depth of the first and second steps will be 30 cm and 40 cm, respectively) . Participants will be asked to stand on the floor confronting the stairs and 20 cm away from the edge of the initial step.

   The stair ascent task will be performed barefooted while arms hanged at the side of the body. Patients will start ascending the steps immediately in response to a command, at their normal speed with their affected limb. Investigators aren't going to control the speed of stair ascent, because controlling the timing of stair-stepping can alter the electromyographic signal as shown earlier for gait in asymptomatic subjects. Before data acquisition, participants will be asked to perform one practice trial of stair ascent to get familiarized with the task. Then the participants will perform three test trials with thirty seconds of rest after each trial to prevent fatigue. The raw data will be stored on a personal computer for analysis with a custom program in Matlab (Math Works, Natick, Massachusetts, USA). Investigators will use a mean of data in three trials for analysis. b) Procedures for treatment: All patients will receive a traditional physical therapy program in the form of TENS , stretching hamstring, quadriceps and calf muscles

   - Group (A) Patients in this group will receive a traditional therapeutic knee rehabilitation program based on a recent systematic review in the form of mini-squatting exercise (up to 45O knee flexion measured by a universal goniometer) , strengthening of hip abductors and external rotators using clamshell exercise . No emphasis will be placed on stabilizing the core musculature before initiating any of those exercises.

   To increase the intensity of exercise, elastic resistance bands will be used.

   - Group (B) Patients in this group will receive the same program as group (A) plus core stability exercise and the principles of core stability will be explained to patients before initiation of treatment and patients will be asked to comply with these principles during exercise. These principles include learning how to activate transversus abdominus by abdominal bracing without allowing pelvis tilting and ensure neutral spine and diaphragmatic breathing during exercise.

   c) Statistical Analysis: Data management and analysis will be conducted using the statistical package for social studies (SPSS) version 22 for windows (IBM SPSS, Chicago, IL, USA). Investigators will conduct the 2X2 Mixed Design MANOVA test to compare the onset and duration of each muscle, pain intensity, and performance of functional activities between group A (traditional therapeutic knee rehabilitation) and group B (core stability) pre-treatment and post-treatment.

ELIGIBILITY:
Inclusion Criteria: patients included if they had

1. Anterior- or retro-patellar knee pain aggravated by at least two activities that load the PFJ (eg; stair ambulation, squatting and/or rising from sitting) .
2. Pain during these activities presented on most days during the past month and their pain severity was ≥ 4 on an 11 point numerical pain scale during aggravating activities .,
3. A grade less than (2) from postero-anterior views on the Kellgren - Lawrence (KL) grading scale.

Exclusion Criteria:

1. concomitant pain from tibiofemoral joint or other knee structures .
2. current or previous pain in the hip, lumbar spine or foot that had lasted longer than 3 months and/or required intervention.
3. a history of lower extremity, pelvis or spine fractures; spine, hip, knee or foot surgeries; hip or patellar subluxation/ dislocation.
4. injury to any of knee ligaments or meniscus.
5. systemic diseases (e.g. rheumatoid arthritis), neurological conditions or fibromyalgia .
6. The professional athletes; people who exercise more than two hours a day or every other day, will be excluded.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
The change of EMG onset of multifidus, | baseline and six weeks
  investigators will collect the EMG activity of multifidus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of multifidus, | baseline and six weeks
  investigators will collect the EMG activity of multifidus using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of transversus abdominus (TrA) muscle | baseline and six weeks
  investigators will collect the EMG activity of TrA using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of transversus abdominus (TrA) muscle | baseline and six weeks
  investigators will collect the EMG activity of TrA using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of gluteus medius (GM) muscle | baseline and six weeks
  investigators will collect the EMG activity of GM using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of gluteus medius (GM) muscle | baseline and six weeks
  investigators will collect the EMG activity of GM using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of vastus medialis obliqus (VMO) muscle | baseline and six weeks
  investigators will collect the EMG activity of VMO using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of vastus medialis obliqus (VMO) muscle | baseline and six weeks
  investigators will collect the EMG activity of VMO using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG onset of vastus lateralis (VL) muscle | baseline and six weeks
  investigators will collect the EMG activity of VL using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).
The change of EMG duration of vastus lateralis (VL) muscle | baseline and six weeks
  investigators will collect the EMG activity of VL using bipolar Ag-AgCl disposable surface electrodes (Better signal solution medical supply Co., limited, Zhongshan, China) and eight channels high-resolution wireless bio amplifier (WBA) system (Biomation, Almonte, Canada).

SECONDARY OUTCOMES:
pain intensity | baseline and six weeks
  The eleven-point numerical rating scale will be used to measure pain severity for patients.where the endpoints are the extremes of no pain and pain as bad as it could be or worst pain. increasing the value means more intense pain.
performance of functional activities | baseline and six weeks
  kujala scale will be used to evaluate the performance of functional activities. This questionnaire includes 13 questions and the scores range from 0 to 100, where 100 indicates the highest efficiency of the knee and 0 indicates the highest disability.

CONTACTS AND LOCATIONS:
Overall Officials: Aladdin A. balbaa, professor, Study Director — Cairo University
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No